CLINICAL TRIAL: NCT05620706
Title: Study of GPC-3 CAR-T Cells in Advanced Hepatocellular Carcinoma
Brief Title: Study of GPC-3 CAR-T Cells in Treating With Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-023
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): GCP3 CAR-T cells
  Interventions: Biological: GPC3 CAR-T cells

INTERVENTIONS:
Biological: GPC3 CAR-T cells — patients treated with GPC3 CAR-T cells

SUMMARY:
Hepatocellular carcinoma is a highly heterogeneous disease. Treatment strategies for advanced hepatocellular carcinoma are limited. Phosphatidylinositol proteoglycan 3 (GPC3) is a heparan sulfate glycoprotein (HSPG) on the surface of the cell membrane. It is highly expressed in liver cancer tissues, but hardly expressed in normal liver tissues. It is an ideal target for tumor treatment. Investigators aimed to test the safety and efficacy of GPC3 CAR-T cells in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is a highly heterogeneous disease. Treatment strategies for advanced hepatocellular carcinoma are limited. Resulting in a poor prognosis. Phosphatidylinositol proteoglycan 3 (GPC3) is a heparan sulfate glycoprotein (HSPG) on the surface of the cell membrane. It is highly expressed in liver cancer tissues, but hardly expressed in normal liver tissues. It is an ideal target for tumor treatment. Investigators aimed to test the safety and efficacy of GPC3 CAR-T cells in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 40~70 years old;
2. Patients with advanced hepatocellular carcinoma (HCC) diagnosed by histopathology or cytology, who are not suitable for surgery or local treatment (including ablation therapy, interventional therapy and radiotherapy), and who have experienced progress or intolerance after receiving standard treatment in the past;
3. Patients who have been terminated for more than 28 days due to previous ineffective PD-1 monoclonal antibody treatment;
4. At least one target lesion that can be evaluated stably according to RECIST 1.1 standard is defined as: the longest diameter of non lymph node lesions ≥ 10mm, or the short diameter of lymph node lesions ≥ 15mm; Intrahepatic lesions require enhanced imaging in arterial phase;
5. Tumor tissue samples were positive for GPC3 by immunohistochemistry (IHC);
6. Grade C according to Barcelona liver cancer grading standard (BCLC) or Grade B which is not suitable for local treatment/progression of local treatment;
7. Estimated survival time > 12 weeks;
8. Cirrhotic state Child Pugh score Grade A
9. ECOG physical status score 0~1;
10. If the patient is HBsAg positive or HBcAb positive, HBV-DNA<200IU/ml. HBsAg positive patients must receive antiviral treatment according to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015);
11. Single vein access;
12. Blood routine test: WBC ≥ 2.5 × 109/L， PLT≥60 × 109/L， Hb≥9.0 g/dL，LY≥0.4 × 109/L；
13. Blood biochemistry: serum Alb ≥ 30 g/L, serum lipase and amylase ≤ 1.5 ULN, serum creatinine ≤ 1.5 ULN and endogenous creatinine clearance rate ≥ 40mL/min, ALT ≤ 5ULN, AST ≤ 5ULN, total bilirubin ≤ 2.5ULN, prothrombin time extension ≤ 4s;
14. The women of childbearing age must carry out serum pregnancy test within the screening period and 14 days before starting the study medication, and the result is negative. They are willing to use reliable methods of contraception during the test period (within 12 months (M12) after cell infusion); For male subjects whose partners are women of childbearing age, they should have undergone sterilization or agree to use reliable methods of contraception during the trial
15. Be able to understand and sign the informed consent form

HBsAg positive patients must receive antiviral treatment according to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015);

11. Single vein access;

12. Blood routine test: WBC ≥ 2.5 × 109/L， PLT≥60 × 109/L， Hb≥9.0 g/dL，LY≥0.4 × 109/L；

13. Blood biochemistry: serum Alb ≥ 30 g/L, serum lipase and amylase ≤ 1.5 ULN, serum creatinine ≤ 1.5 ULN and endogenous creatinine clearance rate ≥ 40mL/min, ALT ≤ 5ULN, AST ≤ 5ULN, total bilirubin ≤ 2.5ULN, prothrombin time extension ≤ 4s;

14. The women of childbearing age must carry out serum pregnancy test within the screening period and 14 days before starting the study medication, and the result is negative. They are willing to use reliable methods of contraception during the test period (within 12 months (M12) after cell infusion); For male subjects whose partners are women of childbearing age, they should have undergone sterilization or agree to use reliable methods of contraception during the trial

15. Be able to understand and sign the informed consent form

Exclusion Criteria:

1. Pregnant or lactating women;
2. HCV-RNA, HIV antibody or syphilis antibody are positive;
3. Any uncontrollable active infection, including but not limited to active tuberculosis;
4. Have received systemic steroids equivalent to>15 mg prednisone within 2 weeks before single collection, except inhaled steroids;
5. Allergies to immunotherapy and related drugs, previous severe allergies β- Allergy to lactam antibiotics;
6. Previous or current hepatic encephalopathy;
7. At present, there is ascites with clinical significance, which is defined as: ascites with positive signs on physical examination or ascites that need to be controlled by intervention (such as puncture or drug therapy) (only those with ascites shown on imaging without intervention can be included);
8. Imaging examination results: the proportion of liver being replaced by tumor ≥ 50%, or portal trunk tumor thrombus, or tumor thrombus invading mesenteric vein/inferior vena cava;
9. Central nervous system metastasis and diseases of central nervous system with clinical significance;
10. At present, there is a heart disease that needs treatment or hypertension that is judged by the researcher to be poorly controlled (systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg);
11. Patients with known active autoimmune diseases need to be treated with immunosuppressants including biological agents;
12. Patients with a history of organ transplantation or waiting for organ transplantation (including liver transplantation);
13. Have received treatment for the study disease within 2 weeks before single collection, including but not limited to surgical treatment, interventional treatment, radiotherapy, chemotherapy and immunotherapy;
14. Received targeted GPC3 treatment, TCR-T treatment and CAR-T treatment in the past month;
15. Being treated with anti PD-1/PD-L1 monoclonal antibody in the past 28 days;
16. Other incurable malignant tumors in the past 5 years or at the same time, excluding cervical carcinoma in situ and skin basal cell carcinoma;
17. Other serious diseases that may restrict the subjects from participating in this trial (such as diabetes under poor control (HbA1c>7% after treatment), severe cardiac insufficiency (LVEF<45%), myocardial infarction or unstable arrhythmia or unstable angina pectoris in the last 6 months, pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease Pulmonary function test FEV1 accounts for less than 60% of the estimated value, gastric ulcer, history of gastrointestinal bleeding disease or clear gastrointestinal bleeding tendency);
18. The investigator assessed that the patient was unable or unwilling to comply with the requirements of the study protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
AE/SAE | from cell infusion to 30 days after infusion
  adverse event/sever adverse event

SECONDARY OUTCOMES:
ORR | From admission to the end of follow up, up to 2 years.
  overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No